CLINICAL TRIAL: NCT01482442
Title: A Prospective Randomized Open-labeled Trial Comparing RADIOEMBOLIZATION With Yttrium 90 Microspheres and Sorafenib in Patients With Advanced Hepatocellular Carcinoma
Brief Title: SorAfenib Versus RADIOEMBOLIZATION in Advanced Hepatocellular Carcinoma
Acronym: SARAH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P101103
Record Dates: First submitted 2011-11-28; First posted 2011-11-30 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2017-01

CONDITIONS: Liver Carcinoma
Keywords: Liver, HCC; Liver, interventional procedures; Liver, randomized studies; Liver, targeted therapy; Liver, RADIOEMBOLIZATION
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sorafenib group (Active Comparator): Patients will receive continuous oral treatment with 800 mg of sorafenib daily (Nexavar, Bayer HealthCare Pharmaceuticals-Onyx Pharmaceuticals). Treatment interruptions and dose reductions (to 400 mg once daily) will be permitted for drug-related adverse effects. At the discretion of the investigator, the dose may be re-escalated to after the resolution of the adverse event.
  Interventions: Drug: sorafenib
- radioembolization group (Active Comparator): The first step will check patient eligibility and prepare conditioning by performing selective mesenteric and hepatic angiography (to document the arterial tumor supply and to occlude extrahepatic vessels) and 99mTc-macroaggregated albumin scintigraphy. The second step is RADIOEMBOLIZATION therapy. One to two weeks after patient eligibility and conditioning, treatment is performed with SIR-Sphere (SIRTEX Medical Ltd.,Lane Cove,Australia).
  Interventions: Drug: SIR-Sphere

INTERVENTIONS:
Drug: sorafenib — Patients will receive continuous oral treatment with 800 mg of sorafenib daily (Nexavar, Bayer HealthCare Pharmaceuticals-Onyx Pharmaceuticals). Treatment interruptions and dose reductions (to 400 mg once daily) will be permitted for drug-related adverse effects. At the discretion of the investigator, the dose may be re-escalated to after the resolution of the adverse event.
  Arms: sorafenib group
Drug: SIR-Sphere — The first step will check patient eligibility and prepare conditioning by performing selective mesenteric and hepatic angiography (to document the arterial tumor supply and to occlude extrahepatic vessels) and 99mTc-macroaggregated albumin scintigraphy. The second step is RADIOEMBOLIZATION therapy. One to two weeks after patient eligibility and conditioning, treatment is performed with SIR-Sphere (SIRTEX Medical Ltd.,Lane Cove,Australia).
  Arms: radioembolization group

SUMMARY:
The purpose of this study is to determine whether RADIOEMBOLIZATION with 90 Yttrium microspheres is more effective on overall survival in advanced Hepatocellular carcinoma (HCC) with or without portal venous obstruction and no extrahepatic extension than sorafenib which is now the standard treatment of advanced HCC.

DETAILED DESCRIPTION:
Background: In patients with advanced hepatocellular carcinoma, sorafenib is now the standard treatment with an increased median overall survival but an overall incidence of treatment-related adverse events of 80%. There is growing interest for RADIOEMBOLIZAION with 90 Yttrium microspheres. It involves infusion of embolic microparticles of glass or resin impregnated with the isotope yttrium-90 through a catheter directly into the hepatic arteries. A substantial number of open-label single-group studies showed supporting evidence for a potential efficacy on overall survival and acceptable or low toxicity. Trial design: multicenter, prospective, controlled, open label randomized trial of Y90 RADIOEMBOLIZATION versus sorafenib. Participants: Adult patients with 1) advanced HCC according to BCLC staging system (stage C) with or without portal vein thrombosis 2) ECOG performance status of 2 or less 3) adequate haematological, renal and hepatic functions 4) liver cirrhosis Child Pugh A - B7 and 5) no extrahepatic metastasis. Interventions: In the sorafenib group, patients will receive continuous oral treatment with 400 mg of sorafenib twice daily. In the Y90 RADIOEMBOLIZATION group, patients will first undergo angiography and scintigraphy for eligibility assessment (absence of or acceptable lung shunting) and preconditioning (embolization). RADIOEMBOLIZATION therapy with infusion of Y90 microspheres will be performed secondly. Objectives: The primary objective is to compare the efficacy of Y90 RADIOEMBOLIZATION to sorafenib in the treatment of advanced hepatocellular carcinoma. Secondary objectives include the comparison of safety profiles, quality of life and health care costs between the two therapeutic groups. Outcomes: The primary endpoint is the median overall survival time. Secondary endpoints include adverse events reported according to the NCI CTC, progression-free survival at 6 months, response rates, general and hepatic-specific quality of life scores, health care costs which comprise the MICROCOSTING of Y90 RADIOEMBOLIZATION from the viewpoint of the hospital and the full cost of each strategy. Sample size: 400 participants (200 par arm). The trial have 80% power to detect a clinically meaningful increase in median survival time of 4 months between sorafenib (expected median survival time 10.7 months) and Y90 RADIOEMBOLIZATION (expected median survival time 15 months) with a two-tailed type I error risk of 5%. Randomization: 1 to 1 randomization will be stratified according to recruiting center, ECOG performance status (a score of 0 vs. a score of 1 or 2), presence or absence of macroscopic vascular invasion (obstruction of portal vein or any branch vs none) and previous chemoembolisation failure . Randomly permuted blocks of random sizes will be used. Study duration and Setting: Accrual period 24 months. Additional follow-up period: 12 months. 14 centres involving both clinicians (hepatologists, hepatobiliary surgeons, and oncologists) and radiologists and Nuclear medicine physicians on each site.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis or meet the AASLD criteria for diagnosis of HCC and at least one uni-dimensional lesion measurable according to RECIST criteria by CT-scan or MRI
* Adult over 18 years old and estimated life expectancy over 3 months
* Patient with advanced HCC according to BCLC staging system (stage C) with or without portal vein thrombosis, not eligible for surgical resection, liver transplantation nor radiofrequency ablation OR patient with progression or recurrence of HCC after surgical or locoregional treatment not eligible for surgical resection, liver transplantation nor radiofrequency ablation OR patients in whom chemoembolisation has failed after two courses (patients who have received only one course of chemoembolisation are eligible if the failure of the first round shows that a second round will have no more impact; patients who have received more than two courses of chemoembolisation are still eligible if the arterial network is perfectly normal on a CT scan in the arterial phase). Failure is defined as the absence of an objective response after two courses of treatment in the treated nodule (objective response according to modified RECIST criteria and/or EASL criteria).
* ECOG performance status under or equals 1
* Adequate haematological function: Hb over or equals 9g/100mL, absolute neutrophil count over or equals 1 500/mm3, platelet count over or equals 50 000/mm3
* Adequate renal function; serum creatinine under 150μmol/L
* Bilirubin under or equals 50 µmol/L, AST or ALT uner or equals 5 x ULN, INR under or equals 1.5
* Liver cirrhosis Child Pugh A - B7
* written informed consent

Exclusion Criteria:

* Another primary tumour, with the exception of conventional basal cell carcinoma or superficial bladder neoplasia
* Extrahepatic metastasis
* Advanced HCC previously treated
* Advanced liver disease with Child-Pugh score over 7 or active gastrointestinal bleeding or encephalopathy or ascites refractory to diuretic therapy Women who are pregnant or breast feeding
* Allergy to contrast media
* Contraindication to hepatic artery catheterisation, such as severe peripheral vascular disease precluding catheterisation
* Psychiatric or other disorder likely to impact on informed consent
* Patient unable and/or unwilling to comply with treatment and study instructions
* Patient unable to swallow oral medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 496 (Actual)
Dates: Start 2011-12; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Median overall survival time | 36 months
  Median overall survival time since randomisation

SECONDARY OUTCOMES:
Common Terminology Criteria for Adverse Events | 36 months
  Adverse events reported according to the National Cancer Institute Common Terminology Criteria for Adverse Events Version 3.0
Progression-free survival | month 6
  Progression-free survival at 6 months
Response rate | 36 months
  Response rate (complete response, partial response, stable disease)
General and hepatic specific quality of life scores | 36 months
  General and hepatic specific quality of life scores
Health care costs | 36 months
  Health care costs which comprise 2 parts: 1) the microcosting of Y90 radioembolization from the viewpoint of the hospital and 2) the full cost of each strategy

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Vilgrain, PD, PhD, Principal Investigator — Department of radiology
Locations (26):
- France (26):
  - CHU Amiens #2, Amiens, Amiens
  - CHU Angers #3, Angers, Angers
  - CHRU Besançon Hôpital Jean Minjoz #21, Besançon, Besançon
  - Hôpital Jean Verdier #25, Bondy, Bondy
  - Hôpital Côte de Nacre #4, Caen, Caen
  - Hôpital Antoine Béclère #29, Clamart, Clamart
  - Hopital beaujon #1, Clichy, Clichy
  - Henri Mondor #24, Créteil, Créteil
  - CHU Dijon Hôpital Bocage #22, Dijon, Dijon
  - CHU Grenoble #5, Grenoble, Grenoble
  - Hôpital Edouard Herriot #6, Lyon, Lyon
  - Lyon La croix Rousse #27, Lyon, Lyon
  - Institut Paoli Calmettes #7, Marseille, Marseille
  - CHU Marseille Hôpital La Timone #23, Marseille, Marseille
  - Hôpital Saint Eloi #8, Montpellier, Montpellier
  - Hôpital de Brabois #9, Nancy, Nancy
  - Hotel Dieu #10, Nantes, Nantes
  - Hôpital de L'Archet #11, Nice, Nice
  - Hôpital Européen Georges Pompidou #13, Paris, Paris
  - Hôpital Haut Leveque #14, Pessac, Pessac
  - CHU Poitiers La Milétrie, Poitiers, Poitiers
  - CHU Robert Debré #28, Reims, Reims
  - CHU Saint Etienne Hôpital Nord #17, Saint-Priest-en-Jarez, Saint-Priest En Jarez
  - Hôpital de Hautepierre #18, Strasbourg, Strasbourg
  - Paul Brousse #19, Villejuif, Villejuif
  - Institut Gustave Roussy #20, Villejuif, Villejuif

REFERENCES:
- [Derived] Zarca K, Mimouni M, Pereira H, Chatellier G, Vilgrain V, Durand-Zaleski I; SARAH Trial Group. Cost-Utility Analysis of Transarterial Radioembolization With Yttrium-90 Resin Microspheres Compared With Sorafenib in Locally Advanced and Inoperable Hepatocellular Carcinoma. Clin Ther. 2021 Jul;43(7):1201-1212. doi: 10.1016/j.clinthera.2021.04.018. Epub 2021 May 28. PMID 34059326
- [Derived] Hermann AL, Dieudonne A, Ronot M, Sanchez M, Pereira H, Chatellier G, Garin E, Castera L, Lebtahi R, Vilgrain V; SARAH Trial Group. Relationship of Tumor Radiation-absorbed Dose to Survival and Response in Hepatocellular Carcinoma Treated with Transarterial Radioembolization with 90Y in the SARAH Study. Radiology. 2020 Sep;296(3):673-684. doi: 10.1148/radiol.2020191606. Epub 2020 Jun 30. PMID 32602828
- [Derived] Vilgrain V, Pereira H, Assenat E, Guiu B, Ilonca AD, Pageaux GP, Sibert A, Bouattour M, Lebtahi R, Allaham W, Barraud H, Laurent V, Mathias E, Bronowicki JP, Tasu JP, Perdrisot R, Silvain C, Gerolami R, Mundler O, Seitz JF, Vidal V, Aube C, Oberti F, Couturier O, Brenot-Rossi I, Raoul JL, Sarran A, Costentin C, Itti E, Luciani A, Adam R, Lewin M, Samuel D, Ronot M, Dinut A, Castera L, Chatellier G; SARAH Trial Group. Efficacy and safety of selective internal radiotherapy with yttrium-90 resin microspheres compared with sorafenib in locally advanced and inoperable hepatocellular carcinoma (SARAH): an open-label randomised controlled phase 3 trial. Lancet Oncol. 2017 Dec;18(12):1624-1636. doi: 10.1016/S1470-2045(17)30683-6. Epub 2017 Oct 26. PMID 29107679
- [Derived] Vilgrain V, Abdel-Rehim M, Sibert A, Ronot M, Lebtahi R, Castera L, Chatellier G; SARAH Trial Group. Radioembolisation with yttrium-90 microspheres versus sorafenib for treatment of advanced hepatocellular carcinoma (SARAH): study protocol for a randomised controlled trial. Trials. 2014 Dec 3;15:474. doi: 10.1186/1745-6215-15-474. PMID 25472660